CLINICAL TRIAL: NCT04088318
Title: A Phase II Study to Evaluate the Safety and Efficacy of OQL011 on VEGFR Inhibitor-Associated Hand-Foot Skin Reaction in Cancer Patients
Brief Title: A Study to Investigate OQL011 on VEGFR Inhibitor-Associated Hand-Foot Skin Reaction in Cancer Patients
Acronym: NOVA-II
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: OnQuality Pharmaceuticals (USA) LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: OQL011B002
Record Dates: First submitted 2019-08-30; First posted 2019-09-12 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2023-09

CONDITIONS: Hand-Foot Skin Reaction (HFSR)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- OQL011 Dose I (Experimental): OQL011, Dose I, ointment, to be applied topically, three times a day, for up to six weeks (in Part 1) or four weeks (in Part 2)
  Interventions: Drug: OQL011
- OQL011 Dose II (Experimental): OQL011, Dose II, ointment, to be applied topically, three times a day, for up to six weeks (in Part 1) or four weeks (in Part 2)
  Interventions: Drug: OQL011
- OQL011 Dose III (Experimental): OQL011, Dose III, ointment, to be applied topically, three times a day, for up to six weeks (in Part 1) or four weeks (in Part 2)
  Interventions: Drug: OQL011
- Vehicle Ointment (Other): Vehicle ointment, to be applied topically, three times a day, for up to six weeks (in Part 1) or four weeks (in Part 2)
  Interventions: Drug: Vehicle Ointment

INTERVENTIONS:
Drug: OQL011 — OQL011 is an ointment containing active ingredient.
  Arms: OQL011 Dose I; OQL011 Dose II; OQL011 Dose III
Drug: Vehicle Ointment — Vehicle ointment is an ointment containing no active ingredient.
  Arms: Vehicle Ointment

SUMMARY:
Hand-Foot Skin Reaction (HFSR) is a common adverse event induced by Vascular Endothelial Growth Receptor Inhibitor (VEGFRi) treatment in cancer patients. The main purpose of this study is to evaluate the safety and efficacy of OQL011 compared to vehicle ointment in treating patients with moderate to severe VEGFRi-associated HFSR. This study will also identify an optimal dosage for Phase III study and explore the pharmacokinetics profile of OQL011 in HFSR patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be age ≥ 18 years.
* Patient must have a confirmed cancer diagnosis for which VEGFRi treatment is indicated, and must be currently under VEGFRi-based anti-cancer therapy with stable dosage for ≥ 1 week. This treatment may be VEGFRi monotherapy or VEGFRi-based combination therapy, so long as it does not include prohibited therapies.
* Patient must have shown signs of HFSR that meet (for Part 1) the NCI CTCAE v5.0 - PPE grade 2 or higher OR (for Part 2) IGA-HFSR criteria of grade 3 or higher.
* Patient on pain medications is allowed provided they have been on stable dosage in the past 1 week and is going to continue at the same dosage.
* Patient is able to use topical medications and complete questionnaires reliably.
* Eastern Cooperative Oncology Group (ECOG) performance score ≤ 2.
* Patient must have the ability to understand and the willingness to sign a written informed consent prior to study entry.

Exclusion Criteria:

* Patient with unresolved hand or foot skin disorders (NCI CTCAE v5.0 grade 2 or higher) due to other medications within 4 weeks prior to study entry.
* Patient who is using other topical medications in the hands or feet area and cannot stop such usage >7 days ahead of randomization.
* Patient who is using other concurrent cancer medications, such as capecitabine, pegylated liposomal doxorubicin, 5-fluorouracil, dabrafenib, vemurafenib, doxorubicin, docetaxel, cytarabine, ramucirumab and bevacizumab, which may result in hand-foot syndrome (HFS).
* Patient who is under uncontrolled intercurrent illness including, but not limited to, inadequately controlled nausea, vomiting, diarrhea or other conditions which may contribute to hypovolemia, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, recent myocardial infarction, uncontrolled hypotension or hypertension, cardiac arrhythmia, or psychiatric illness and social situations that would limit compliance with study requirements.
* Patient who has contraindication with the active compound, including severe anemia, increased intracranial pressure, known hypersensitivity.
* Patient who has other skin disorders that will affect the efficacy evaluation on hands and feet area, including but not limited to, tinea of feet and hands, hand/foot eczema, palmoplantar pustulosis, palmoplantar keratosis, acrodermatitis continua etc.
* Patient who used phosphodiesterase type 5 (PDE5) inhibitors such as sildenafil, vardenafil, and tadalafil within past 7 days.
* Patient with significantly abnormal lab test:

  * Inadequate hematologic function as indicated by:

    * Absolute neutrophil counts (ANC) ≤ 1,000 /mm^3
    * Hemoglobin (Hgb) ≤ 8.0 g/dL
    * Platelet count ≤ 75,000 /mm^3
    * PT or PTT > 1.5 x ULN (if patients on anticoagulants: PT INR > 3.5 x ULN)
  * Inadequate renal and liver function as indicated by:

    * Albumin < 2.8 g/dL
    * Total bilirubin ≥ 1.5 x ULN (or ≥ 2.5 x ULN for patients with Gilbert's syndrome)
    * Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase ≥ 3 x ULN (or ≥ 5 x ULN for patients with liver cancer)
    * Creatinine > 2.0 x ULN.
* Pregnant or nursing women.
* Women of childbearing potential who are unwilling to comply with contraceptive requirements. Highly effective contraception which include two forms of birth control method (i.e., a hormonal method plus a barrier method) is advised for at least 2 weeks prior to study treatment and during study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2019-12-09 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
(For Part 1) Proportion of patients who achieve NCI CTCAE v5.0 - Palmar-Plantar Erythrodysesthesia (PPE) grade 0 or 1 OR (for Part 2) The proportion of patients achieving IGA-HFSR grade 0 or 1 | 3 weeks (Part 1) OR 2 weeks (Part 2)

SECONDARY OUTCOMES:
(For Part 1) Proportion of patients who have improvement in HFSR severity and achieve clear (0) or almost clear (1) as measured by IGA-i (Investigator-assessed Investigator's Global Assessment) scale | 3 weeks and 6 weeks
  The IGA scale ranges from grade 0 (clear) to 4 (severe), the higher the score, the worse the condition.
(For Part 2) Proportion of patients achieving IGA-HFSR grade 0 or 1 | 4 weeks
  The IGA scale ranges from grade 0 (clear) to 4 (severe), the higher the score, the worse the condition.
(For Part 2) Proportion of patients achieving at least two-grade improvement in IGA-HFSR | 2 weeks and 4 weeks
  The IGA scale ranges from grade 0 (clear) to 4 (severe), the higher the score, the worse the condition.
(For Part 1) Proportion of patients who achieve NCI CTCAE v5.0 - PPE grade 0 or 1 | 6 weeks
(For Part 2) Change from baseline in NCI CTCAE v5.0 - PPE grade | 2 weeks and 4 weeks
Change from baseline in HF-QoL (Hand-Foot Skin Reaction and Quality of Life) Questionnaire total score | 3 weeks and 6 weeks (Part 1) OR 2 weeks and 4 weeks (Part 2)
  HF-QoL questionnaire is comprised of a 20-item symptom domain and an 18-item daily activity domain. Each item is rated on a 5-point scale from 0 (not at all) to 4 (always or extremely) during the previous week. The HF-QoL symptom and daily activity total scores are transformed to a scale of 0 to 100, based on the sum of each unit-weighted item score divided by the maximum score. Higher scores on the HF-QoL indicate worse quality of life or greater symptom burden. (refer to R. T. Anderson et al., The Oncologist 2015;20:831-838)
(For Part 1) Change from baseline in patient reported pain using VAS (Visual Analog Scale) | 3 weeks and 6 weeks
  The subject records pain associated with HFSR using 100 mm VAS ranging from "no pain" at 0 mm to "unbearable pain" at 100 mm on the paper VAS.
(For Part 2) Change from baseline in patient reported pain using NPRS (Numerical Pain Rating Scale) | 2 weeks and 4 weeks
  The subject records pain associated with HFSR using score 0 to 10 ranging from "no pain" for Score 0 to "unbearable pain" for Score 10.
(For Part 1) Proportion of patients who have improvement in HFSR severity and achieve clear (0) or almost clear (1) as measured by IGA-c (Centrally-assessed Investigator's Global Assessment) scale | 3 weeks and 6 weeks
  The IGA scale ranges from grade 0 (clear) to 4 (severe), the higher the score, the worse the condition.
Safety assessment by type, incidence and intensity of adverse events | 6 weeks (Part 1) and 4 weeks (Part 2)
Plasma concentration of active compound and its derivatives | 1 day
(For Part 2) The exposure-response relationship of different dose level OQL011 | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mario E. Lacouture, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (33):
- United States (15):
  - Western Regional Medical Center, Goodyear, Arizona
  - Innovative Clinical Research Institute, Whittier, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Yale University - Hospital, New Haven, Connecticut
  - AP Medical Research, Miami, Florida
  - Northwestern University - Hospital, Chicago, Illinois
  - University of Louisville - Hospital, Louisville, Kentucky
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Innovative Clinical Research Institute, Henderson, Nevada
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Montefiore Einstein Center for Cancer Care, The Bronx, New York
  - Gabrail Cancer Centre, Canton, Ohio
  - Ohio State University Dermatology, Columbus, Ohio
  - MD Anderson Cancer Center, Houston, Texas
- China (10):
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - Taizhou People's Hospital, Taizhou, Jiangsu
  - Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Tongren Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
- India (8):
  - S.P Medical College & AG Hospitals, Bikaner, Bīkaner, Dimhans
  - Kiran Multi Super Speciality Hospital & Research Center, Surat, Gujarat
  - Kailash Cancer Hospital and Research Center, Vadodara, Gujarat
  - Aadhar Health Institute, Hisar, Haryana
  - Noble Hospital, Pune, Hisar, Haryana
  - Oncoville Cancer Hospital and Research Center, Bangalore, Karnataka
  - Mumbai Oncocare Centre, Mumbai, Maharashtra
  - HCG Manavata Cancer centre, Nashik, Nāka, Nashik

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.